CLINICAL TRIAL: NCT05529784
Title: Effectiveness of Dupilumab in the Treatment of Severe Uncontrolled CRSwNP: a Multicentre Observational Real-life Study (DUPIREAL)
Brief Title: Dupilumab in the Treatment of Severe Uncontrolled CRSwNP: a Multicentre Observational Real-life Study (DUPIREAL)
Acronym: DUPIREAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DE CORSO EUGENIO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0034704/21
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe, uncontrolled CRSwNP patients in therapy with Dupilumab
  Interventions: Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]

INTERVENTIONS:
Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT] — Dupilumab 300mg in pre-filled injector Q2W

SUMMARY:
Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) is a sino-nasal chronic inflammatory disease that strongly affects patients' quality of life, especially in difficult-to-treat cases. In severe uncontrolled CRSwNP, the inflammation is mostly driven by a type 2 inflammatory pathway and its management has been rapidly changing during the last 2 years due to Dupilumab approval. It is a fully human monoclonal antibody that binds the alpha subunit of IL-4 receptors (IL-4Rα type 1 and type 2) to inhibit IL-4 and IL-13 signaling.

So far, randomized clinical trials have assessed efficacy and safety of Dupilumab in a large number of patients, whereas evidences in real life clinical practice are limited to few monocentric series.

Herewith, the investigators present a multicenter, observational nationwide retrospective real-life study with the aim to confirm the effectiveness and the safety of Dupilumab over the first year of treatment in a real life setting.

The primary objective is to evaluate the volumetric reduction of polyps by measuring the variation of total Nasal Polyp Endoscopic Score (NPS).

The secondary objectives are:

* the evaluation of changes in nasal symptoms, olfactory function and nasal obstruction
* the assessment of the patients' quality of life
* the recording of major and minor complications
* the evaluation of the response to the therapy, according to EPOS2020 criteria and EUFOREA2021
* the assessment of efficacy based on concomitant disease (Asthma and ASA triad)
* the evaluation of potential predictors of clinical response to the therapy

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of diffuse CRSwNP by endoscopy and CT scan performed at least 6 months prior of the therapy;
* severe disease stage defined by NPS ≥5 or SNOT-22 ≥50;
* inadequate symptom control with INCS therapy;
* failure or intolerance of previous medical treatments (at least 2 cycles of systemic corticosteroid in the last year), and/or failure of previous surgical treatment through nasal endoscopic surgery (ESS), with postoperative complications or no clinical benefit

Exclusion Criteria:

* pregnant women;
* immunosuppressive therapy;
* patients undergoing radio-chemotherapy treatments for cancer in the 12 months before the starting of therapy;
* concomitant long-term corticosteroid therapy for chronic autoimmune disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We included all the patients that were referred to Dupilumab therapy, prescribed accordingly to the plan provided by Italian Agency of Drugs.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score (NPS) | 12 months
  Polyps volume. Range 0-4 for each nostril. Higher score describes a worse condition

SECONDARY OUTCOMES:
Nasal Polyp Score (NPS) | 24 months
  Polyps volume. Range 0-4 for each nostril. Higher score describes a worse condition
Nasal congestion score (NCS) | 12 months and 24 months
  Nasal congestion. Range 0-3. Higher score describes a worse condition
Sinonasal outcome test (SNOT-22) | 12 months and 24 months
  Symptoms. Range 0-110. Higher score describes a worse condition
Sniffin' sticks identification test | 12 months and 24 months
  Olfaction. Range 0-16. Higher score describes a better condition
Visual Analog Scale (VAS) for nasal congestion | 12 months and 24 months
  Nasal congestion. Range 0-10. Higher score describes a more severe symptom
Visual Analog Scale (VAS) for olfaction loss | 12 months and 24 months
  Olfaction loss. Range 0-10. Higher score describes a more severe symptom
Visual Analog Scale (VAS) for craniofacial pain | 12 months and 24 months
  Craniofacial pain. Range 0-10. Higher score describes a more severe symptom
Visual Analog Scale (VAS) for sleeping disorders | 12 months and 24 months
  Sleeping disorders. Range 0-10. Higher score describes a more severe symptom
Visual Analog Scale (VAS) for rhinorrhea | 12 months and 24 months
  Rhinorrhea. Range 0-10. Higher score describes a more severe symptom
Visual Analog Scale (VAS) for quality of life | 12 months and 24 months
  Quality of life. Range 0-10. Higher score describes a worse quality of life
Need for surgery | 12 months and 24 months
  Number of surgeries performed during therapy
Intranasal corticosteroid adherence | 12 months and 24 months
  Number of days of suspension of intranasal corticosteroids
Need for rescue oral corticosteroids | 12 months and 24 months
  Number of short cycles of oral corticosteroids during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio De Corso, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (19):
- Italy (19):
  - AUSL Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Policlinico S. Marco, Catania
  - AUSL Latina, Latina
  - ASST Santi Paolo e Carlo - Presidio San Paolo, Milan
  - IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - A.O.R.N. Ospedali dei Colli, Napoli
  - Azienda Ospedaliera Policlinico Federico II, Napoli
  - Ospedale maggiore di Novara, Novara
  - Ospedale S.Luigi Gonzaga, Università di Torino, Orbassano
  - Azienda Ospedaliero-Universitaria di Padova, Padua
  - Policlinico San Matteo-Università di Pavia, Pavia
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia
  - ASL Roma 5, Roma
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma
  - Università La Sapienza, Roma
  - Azienda Ospedaliero-Universitaria di Sassari, Sassari

IPD SHARING:
Plan to Share IPD: Undecided